CLINICAL TRIAL: NCT00358579
Title: A Randomised, Double-blinded Multi-centre Trial Comparing Vasopressin and Adrenaline in Patients With Cardiac Arrest at the Emergency Department. (Preadmission Intravenous Vasopressin, Adrenaline Outcome Trial: PIVOT vII)
Brief Title: Comparing Vasopressin and Adrenaline in Patients With Cardiac Arrest
Acronym: PIVOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Alexandra Hospital (Other); National University Hospital, Singapore (Other); Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SQCA01
Record Dates: First submitted 2006-07-30; First posted 2006-08-01 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Arrest
Keywords: Vasopressin; Adrenaline; Survival; Return of spontaneous of circulation
MeSH Terms: conditions — Heart Arrest; Diabetes Insipidus | interventions — Epinephrine; Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adrenaline (Active Comparator)
  Interventions: Drug: Adrenaline
- Vasopressin (Active Comparator)
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Adrenaline — 1 mg
  Other Names: Epinephrine
  Arms: Adrenaline
Drug: Vasopressin — 40 IU
  Other Names: Arginine vasopressin; argipressin; antidiuretic hormone
  Arms: Vasopressin

SUMMARY:
The effectiveness of medications in cardiac arrest has been greatly debated and questioned. Historically intravenous adrenaline has been the drug of choice since 1906. There have been few formal evaluations to determine the value of adrenaline for cardiac arrest, and clinical trials have not been able to show any benefit with intravenous adrenaline (compared to placebo or no treatment) in the field.

Thus the purpose of this study is to compare vasopressin and adrenaline in the treatment of cardiac arrest to answer the question whether there is an improvement in survival between vasopressin and adrenaline.

DETAILED DESCRIPTION:
The effectiveness of medications in cardiac arrest has been greatly debated and questioned. Historically intravenous adrenaline has been the recommended drug of choice since 1906. There have been few formal evaluations to determine the value of adrenaline for cardiac arrest, and clinical trials have not been able to show any benefit with intravenous adrenaline (compared to placebo or no treatment) in the field.

More recently, vasopressin has been used in patients with cardiac arrest. In human studies on vasopressin, clinical trials have produced conflicting results.

The current study compared vasopressin and adrenaline in the treatment of cardiac arrest in patients presenting to the Emergency Department (ED). Specific outcomes included return of spontaneous circulation (ROSC) (as measured by the presence of a palpable pulse at any time during resuscitation), survival to hospital admission, survival to discharge from hospital, and functional status at discharge and at one year (as measured by the Glasgow-Pittsburgh outcome categories).

ELIGIBILITY:
Inclusion Criteria:

* Patient with cardiac arrest as confirmed by the absence of a pulse, unresponsiveness and apnea
* Age above 16 (Age 21 and above for CGH only)

Exclusion Criteria:

* Traumatic cardiac arrest
* Age 16 and below (Age 20 and below for CGH only)
* CPR is contraindicated

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2006-03; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus EH Ong, MBBS, Principal Investigator — Singapore General Hospital
Locations (4):
- Singapore (4):
  - National University Hospital, Singapore
  - Alexandra Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore

REFERENCES:
- [Derived] Ong ME, Tiah L, Leong BS, Tan EC, Ong VY, Tan EA, Poh BY, Pek PP, Chen Y. A randomised, double-blind, multi-centre trial comparing vasopressin and adrenaline in patients with cardiac arrest presenting to or in the Emergency Department. Resuscitation. 2012 Aug;83(8):953-60. doi: 10.1016/j.resuscitation.2012.02.005. Epub 2012 Feb 18. PMID 22353644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 9 March 2006 to 19 January 2009. Location of recruitment was in emergency departments.
Pre-assignment Details: The exclusion criteria included traumatic cardiac arrest or when cardiopulmonary resuscitation was contraindicated; for example those 'obviously dead' as defined by the presence of decomposition, rigor mortis or dependant lividity. Participants below the age of 16 years old were not included in the study
Groups:
- Adrenaline: 1 mg Intravenous Adrenaline, administered as the first drug upon cardiac arrest patient's arrival at the Emergency Department
- Vasopressin: 40 IU Intravenous Vasopressin, administered as the first drug upon cardiac arrest patient's arrival at the Emergency Department
Period: Overall Study
Arm/Group | Adrenaline | Vasopressin
Started | 353 | 374
Completed | 353 | 374
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adrenaline | Vasopressin | Total
Number analyzed (Participants) | 353 | 374 | 727
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 170 | 186 | 356
  >=65 years | 182 | 188 | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (15.4) | 64.6 (14.2) | 64.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 111 | 222
  Male | 242 | 263 | 505
Region of Enrollment [Number; unit: participants]
  Singapore | 353 | 374 | 727

OUTCOME MEASURES:

1. Primary Outcome: Survival to Hospital Discharge.
Description: Survival to hospital discharge is defined as the patient leaving the hospital alive or survival to 30 days post cardiac arrest,whichever came first. This therefore measures the number of participants who was discharged alive or survived to 30 days post cardiac arrest, whichever came first.
Time Frame: at 30 days post arrest
Measure: Number; unit: Participants
Arm/Group | Adrenaline | Vasopressin
Number analyzed (Participants) | 353 | 374
Participants | 8 | 11

2. Secondary Outcome: Neurological Status on Discharge or at 30 Days Post Arrest, if Not Discharged.
Description: Neurological status is assessed by the Glasgow-Pittsburgh outcome categories, to evaluate quality of life after successful resuscitation. Good neurological status is defined as cerebral performance categories(CPC)/overall performance categories(OPC):1 and 2.CPC/OPC 1 indicates good cerebral & overall performance. CPC/OPC 2 indicates moderate cerebral & overall disability. CPC/OPC 3 indicates severe cerebral & overall disability. CPC/OPC 4 indicates coma, vegetative state. CPC/OPC 5 indicates brain dead/death.
Time Frame: at 30 days post arrest
Measure: Number; unit: Participants
Arm/Group | Adrenaline | Vasopressin
Number analyzed (Participants) | 353 | 374
Participants
  Cerebral Performance Categories 1 | 5 | 4
  Cerebral Performance Categories 2 | 0 | 1
  Overall Performance Categories 1 | 2 | 5
  Overall Performance Categories 2 | 3 | 0

3. Secondary Outcome: Neurological Status at 1 Year.
Description: Neurological status is assessed by the Glasgow-Pittsburgh outcome categories, to evaluate quality of life after successful resuscitation. Good neurological status is defined as cerebral performance categories(CPC)/overall performance categories(OPC): 1 and 2. CPC/OPC 1 indicates good cerebral & overall performance. CPC/OPC 2 indicates moderate cerebral & overall disability. CPC/OPC 3 indicates severe cerebral & overall disability. CPC/OPC 4 indicates coma, vegetative state. CPC/OPC 5 indicates brain dead/death.
Time Frame: at 1 year post arrest
Measure: Number; unit: Participants
Arm/Group | Adrenaline | Vasopressin
Number analyzed (Participants) | 353 | 374
Participants
  Cerebral Performance Categories 1 | 5 | 4
  Cerebral Performance Categories 2 | 0 | 1
  Overall Performance Categories 1 | 3 | 3
  Overall Performance Categories 2 | 2 | 1

4. Secondary Outcome: Return of Spontaneous Circulation.
Description: Return of spontaneous circulation is defined as the presence of any palpable pulse detected by manual palpation of a major artery. This is measured as number of participants who had return of spontaneous circulation during resuscitation.
Time Frame: during resuscitation
Measure: Number; unit: Participants
Arm/Group | Adrenaline | Vasopressin
Number analyzed (Participants) | 353 | 374
Participants | 106 | 119

5. Secondary Outcome: Survival to Admission.
Description: Survival to admission is defined as the presence of pulse on admission to hospital (discharged from Emergency Department and admitted to Intensive Care Units /wards). This measures the number of participants with pulse and who were admitted to hospital.
Time Frame: No specific time frame. Survival to admission refers to sustained return of spontaneous circulation until admission and transfer of care to Intensive Care Units /wards
Measure: Number; unit: Participants
Arm/Group | Adrenaline | Vasopressin
Number analyzed (Participants) | 353 | 374
Participants | 59 | 83

ADVERSE EVENTS:
Description: Serious and other adverse events were not collected or assessed as it is not applicable to this study, which recruits patients in cardiac arrest (low survival rate).
Arm/Group | Adrenaline | Vasopressin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
As the study was conducted over a relatively long period, results may be affected by secular trends.Variations in post-resuscitation care can affect survival to discharge status and variations between institutions are difficult to account for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No